CLINICAL TRIAL: NCT04989400
Title: Use of Ulipristal Acetate in Induction of Second Trimester Missed Abortion in Women With Previous Caesarian Section: A Randomized Controlled Trial.
Brief Title: Use of Ulipristal Acetate in Induction of Second Trimester Missed Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Safwat, lecturer of obstetrics and gynaecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5181
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Induction of Second Trimester Abortion
MeSH Terms: interventions — ulipristal acetate; Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ulipristal group (Experimental): received Ulipristal acetate 30mg, starting misoprostol 12 hours later 100µg every 6 hours buccal according to FIGO guidelines 2017,Then women had rest for 24 hours after 5 doses of misoprostol and restarted misoprostol-only in both groups with the same above regimens, repeating the same sequence for two weeks unless there was excessive bleeding or infection or uterine contractions or cervical changes. If failed, patient proceeded to hysterotomy
  Interventions: Drug: Ulipristal Acetate; Drug: Misoprostol
- placebo (Placebo Comparator): received placebo tablet of same shape , texture of that of ulipristal then 12 hours later start misoprostol 100µg every 6 hours buccal according to FIGO guidelines 2017. Then women in had rest for 24 hours after 5 doses of misoprostol and restarted misoprostol-only in both groups with the same above regimens, repeating the same sequence for two weeks unless there was excessive bleeding or infection or uterine contractions or cervical changes. If failed, patient proceeded to hysterotomy
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Ulipristal Acetate — Group A: received Ulipristal acetate 30mg, starting misoprostol 12 hours later 100µg every 6 hours buccal. Then women in had rest for 24 hours after 5 doses of misoprostol and restarted misoprostol-only in both groups with the same above regimens, repeating the same sequence for two weeks unless there was excessive bleeding or infection or uterine contractions or cervical changes. If failed, patient proceeded to hysterotomy. If patient aborted, an obstetric US was done to assess the presence of remnants in the uterine cavity. Patient with remnants of conception proceeded suction evacuation.
  Arms: ulipristal group
Drug: Misoprostol — Group A: received Ulipristal acetate 30mg, starting misoprostol 12 hours later 100µg every 6 hours buccal.Group B: received placebo tablet of same shape , texture of that of ulipristal then 12 hours later start misoprostol 100µg every 6 hours buccal. Then women in both groups had rest for 24 hours after 5 doses of misoprostol and restarted misoprostol-only in both groups with the same above regimens, repeating the same sequence for two weeks unless there was excessive bleeding or infection or uterine contractions or cervical changes. If failed, patient proceeded to hysterotomy. If patient aborted, an obstetric US was done to assess the presence of remnants in the uterine cavity. Patient with remnants of conception proceeded suction evacuation.

SUMMARY:
The aim of this work is to assess the effectiveness and safety of Ulipristal Acetate in the management of 2nd trimester missed abortion along with misoprostol in pregnant women with previous caesarean section versus the use of misoprostol only with placebo as regards the time needed for abortion,Hypothesis: In pregnant women with 2nd trimester missed abortion with previous caesarean section , Ulipristal Acetate may decrease the time interval to achieve abortion when combined with Misoprostol in comparison to misoprostol alone.the included women divided to 2 groups Group A: will receive Ulipristal acetate 30mg, starting misoprostol 12 hours later 100µg every 6 hours buccal according to FIGO guidelines 2017.Group B: will receive placebo then 12 hours later start misoprostol 100µg every 6 hours buccal according to FIGO guidelines 2017. then we assess Induction-to-abortion interval time.

ELIGIBILITY:
Inclusion Criteria: • Women with 2nd trimester missed abortions

* Gestational age 13-26 weeks.
* Women with a previous caesarian section scar,(para 1cs till para 4 cs).
* Women counseled and chose medication abortion rather than surgical evacuation

Exclusion Criteria:

* Women with an accompanying medical disorder such as: Preeclampsia, Diabetes Mellitus or Heart disease.
* Primigravida women or non scarred uterus.
* Women with previous myomectomy or hysterotomy scar or upper segment caesarean section scar.
* Induction of abortion in women with congenital fetal malformations or positive fetal pulsations due to medical disorder.
* Women with placenta previa .
* Allergy or contraindications to either Ulipristal acetate or Misoprostol.
* Women with inevitable abortion in the form of vaginal bleeding or uterine contractions

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Induction-to-abortion interval time. | 2 weeks
  calculate the time needed from start of intervention till abortion occured

SECONDARY OUTCOMES:
complete evacuation between both groups | 2 weeks
  number of patients experienced complete abortion between both groups
need for hysterotomy | 2 weeks
  number of patients underwent hysterotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04989400/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04989400/SAP_001.pdf